CLINICAL TRIAL: NCT01409564
Title: Cilostazol Augmentation Study In Dementia (CASID): A Randomized, Placebo-controlled Pilot Study to Compare the Efficacy Between Donepezil Monotherapy and Cilostazol Augmentation Therapy in Alzheimer's Disease Patients With Subcortical White Matter Hyperintensities
Brief Title: Cilostazol Augmentation Study in Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea OIAA (Unknown)
Responsible Party: Principal Investigator, Jung-Seok Choi, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-2009-145
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Dementia
Keywords: Alzheimer's dementia; Cilostazol
MeSH Terms: conditions — Alzheimer Disease | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cilostazol (Experimental): Cilostazol group means dementia patients group receiving donepezil with cilostazol augmentation.
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator): Placebo group means dementia patients group receiving donepezil with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100mg bid per day will be administered orally and the period is total 24 weeks. The first week is a period for increasing the quantity, and during this period, cilostazol 50mg bid per day will be administered orally.
  Arms: Cilostazol
Drug: Placebo — Placebo with similar shape and color to cilostazol 100mg bid per day will be administered orally and the period is total 24 weeks. The first week is a period for increasing the quantity, and during this period, placebo 50mg bid per day will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of cilostazol augmentation in mild to moderate Alzheimer disease patients with subcortical white matter hyperintensities (WMHI) treated by donepezil.

Dementia is the most disabling disease in the old age. The prevalence of dementia is 5-10% of the elders. AchEIs (donepezil, galantamine, rivastigmine) are used to treat mild to moderate dementia, but these drugs only relate to symptomatic improvement and the response rates are less than 30%.

Cilostazol is a cyclic adenosine monophosphate phosphodiesterase 3 inhibitor (PDE3I) and used as antiplatelet agent in subcortical vascular disease (WMHI). And it upregulates phosphorylation of cyclic adenosine monophosphate-pathway response element binding protein (CREB) which plays a crucial role in memory enhancement and synaptic plasticity related to neurodegeneration prevention.

The investigators will try cilostazol augmentation in dementia patients with WMHI receiving donepezil to see the addictive effects of cilostazol using cognitive tasks and PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* Men/women over sixty years old
* Patients with slight and moderate dementia (MMSE score is over 10 under 26.)
* Patients with probable Alzheimer's disease according to the standard of NINCDS-ADRDA
* Patients accompanied with WMHI on Brain MRI (Fazeka's scale 1~3)

Exclusion Criteria:

* Those who do not agree to the test in a written form
* Patients who accompany other diseases except cerebral atrophy or change of subcortical white matter due to Alzheimer's disease on brain MRI
* Patients who should not use Cilostazol (① patients with bleeding tendency ② patients with congestive heart failure ③ patients who have a medical history of hypersensitivity to this medicine or constituent of this medicine ④ those who use anticoagulant and clot buster)
* Patients who suffer from nerve diseases or mental diseases which have influence on cognitive function except Alzheimer's disease (for example, schizophrenia, severe depression, mental retardation and etc.)
* Patients who are suspected to have a personal history of drug addiction or alcoholism within recent 10 years
* Patients who have severe problems in eye sight or hearing so that it is impossible to conduct the test smoothly
* Patients who the researchers think are inappropriate for taking part in the test

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Seok Choi, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center, Seoul, Republic of Korea
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee JY, Lee H, Yoo HB, Choi JS, Jung HY, Yoon EJ, Kim H, Jung YH, Lee HY, Kim YK. Efficacy of Cilostazol Administration in Alzheimer's Disease Patients with White Matter Lesions: A Positron-Emission Tomography Study. Neurotherapeutics. 2019 Apr;16(2):394-403. doi: 10.1007/s13311-018-00708-x. PMID 30761509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 Subjects were enrolled in the single center of Seoul National University Boramae Hospital. The diagnosis of probable AD was made according to the criteria of NINCDS-ADRDA (MMSE score 10 ~ 26). Enrollment has started in July 2010 to end in March 2012.
Groups:
- Cilostazol: Cilostazol group includes dementia patients receiving donepezil with cilostazol augmentation. All the randomly assigned AD patients in cilostazol group received 10 mg of Donepezil along with 200 mg of cilostazol per a day, doubly blinded. All the medications were orally administered. For the initial two weeks, patients only received 100 mg of cilstazol per a day to minimize the instabilities. Afterwards, for 22 weeks, patients received 200 mg of cilostazol.
- Placebo: Placebo group includes dementia patients receiving donepezil with placebo. All the patients were randomly assigned as placebo group and received 10 mg of Donepezil along with the same dose of sugar pill as normal cilostazol. All the clinical assessments and medications were doubly blinded. All the medications were orally administered.
Period: Overall Study
Arm/Group | Cilostazol | Placebo
Started | 23 | 23
Completed | 18 | 18
Not Completed | 5 | 5
Not completed — low medication compliance | 4 | 3
Not completed — brain abnormalities found in T1 MR | 1 | 2

BASELINE CHARACTERISTICS:
Population: 18 subjects for each group were enrolled in the final list.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.00 (6.26) | 78.05 (6.09) | 78.53 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Regionally Averaged Cerebral Glucose Uptake Changes Measured by FDG PET Uptake With Voxel-based Method
Description: Regional cerebral glucose uptake level was measured as the ratio value of FDG uptake of the each unit level to the global mean uptake value.
Time Frame: Baseline, 24-week
Population: Number of patients with increased whole brain glucose uptake level. In the real analysis, however, a voxel-based image analysis results were used; therefore, data which can be entered here is not much meaningful.
Measure: Mean (Standard Deviation); unit: Bq/Bq (no unit)
Groups:
- Cilostazol, Baseline: Cilostazol group means dementia patients group receiving donepezil with cilostazol augmentation at the baseline.
- Cilostazol, 24-week: Cilostazol group means dementia patients group receiving donepezil with cilostazol augmentation after 24 weeks.
- Placebo, Baseline: Placebo group means dementia patients group receiving donepezil with placebo at the baseline.
- Placebo, 24-week: Placebo group means dementia patients group receiving donepezil with placebo after 24 weeks.
Arm/Group | Cilostazol, Baseline | Cilostazol, 24-week | Placebo, Baseline | Placebo, 24-week
Number analyzed (Participants) | 18 | 18 | 18 | 18
Bq/Bq (no unit)
  Left Parietal Lobe | 81.70 (9.51) | 80.40 (8.27) | 84.60 (7.47) | 81.33 (6.82)
  Right Parietal Lobe | 80.03 (10.26) | 79.00 (9.55) | 85.29 (8.62) | 81.91 (8.37)
  Left Inferior Frontal Gyrus | 85.74 (7.03) | 86.82 (6.06) | 85.97 (5.72) | 83.12 (5.81)
  Right Inferior Frontal Gyrus | 72.11 (6.48) | 71.39 (4.82) | 74.02 (6.38) | 71.44 (5.53)
Statistical Analysis 1: Comparison: Cilostazol, Baseline vs Cilostazol, 24-week vs Placebo, Baseline vs Placebo, 24-week; Repeated-measures analysis of variance (ANOVA) was used to test group*time interaction effect in glucose uptake of Left Parietal Lobe in two groups on two data points (baseline, 24-week); Test type: Superiority or Other; p = 0.14, Repeated ANOVA; Uncorrected, Repeated ANOVA
Statistical Analysis 2: Comparison: Cilostazol, Baseline vs Cilostazol, 24-week vs Placebo, Baseline vs Placebo, 24-week; Repeated-measures analysis of variance (ANOVA) was used to test group*time interaction effect in glucose uptake of Right Parietal Lobe in two groups on two data points (baseline, 24-week); Test type: Superiority or Other; p = 0.08, Repeated ANOVA
Statistical Analysis 3: Comparison: Cilostazol, Baseline vs Cilostazol, 24-week vs Placebo, Baseline vs Placebo, 24-week; Repeated-measures analysis of variance (ANOVA) was used to test group*time interaction effect in glucose uptake of Left Inferior Frontal Gyrus in two groups on two data points (baseline, 24-week); Test type: Superiority or Other; p < 0.01, Repeated ANOVA
Statistical Analysis 4: Comparison: Cilostazol, Baseline vs Cilostazol, 24-week vs Placebo, Baseline vs Placebo, 24-week; Repeated-measures analysis of variance (ANOVA) was used to test group*time interaction effect in glucose uptake of Right Inferior Frontal Gyrus in two groups on two data points (baseline, 24-week); Test type: Superiority or Other; p = 0.08, Repeated ANOVA

2. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog)
Description: The ADAS-Cog score is measured by the number of questions answered incorrectly, therefore the higher is the worse.
  Score Scale: 0-75 (min-MAX)
  Each subcategory scores are summed.
  1. Word-recall test (0-10)
  2. Commands (0-5)
  3. Constructional praxis (0-5)
  4. Naming Objects/ Fingers (0-5)
  5. Ideational Praxis (0-5)
  6. Orientation (0-8)
  7. Word Recognition (0-12)
  8. Remembering Test Instructions (0-5)
  9. Spoken Language Ability (0-5)
  10. Word Finding Difficulty (0-5)
  11. Comprehension (0-5)
Time Frame: Baseline, 12-week, 24-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 29.28 (8.79) | 27.78 (7.89)
  12-week | 26.33 (6.75) | 24.83 (7.67)
  24-week | 25.78 (8.19) | 24.78 (7.41)
Statistical Analysis 1: Comparison: Cilostazol vs Placebo; Repeated ANOVA, tested for group*time interaction effect of ADAS-Cog scores on three data points (Baseline, 12-week, 24-week); Test type: Superiority or Other; p = 0.93, Repeated ANOVA

3. Secondary Outcome: Mini-Mental State Examination (MMSE) in the Korean Version of the CERAD Assessment Packet)
Description: Basic cognitive functions are checked. (0-30) The score is better when higher.
Time Frame: Baseline, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 15.11 (3.61) | 15.44 (3.96)
  12-week | 16.67 (4.04) | 15.83 (4.84)
  24-week | 15.39 (3.94) | 16.22 (4.91)
Statistical Analysis 1: Comparison: Cilostazol vs Placebo; Repeated ANOVA, tested for group*time interaction effect of MMSE scores on three data points (Baseline, 12-week, 24-week); Test type: Superiority or Other; p = 0.15, Repeated ANOVA

4. Secondary Outcome: Activities of Daily Living (ADCS-ADL)
Description: The caregiver answered to the questions given to measure the cognitive function level of the patients in daily living. Lower scores indicate greater severity.
  23 questions Score Scale: 0-78 (min-MAX)
Time Frame: Baseline, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 50.17 (11.61) | 53.56 (14.86)
  12-week | 48.00 (13.14) | 49.33 (17.38)
  24-week | 46.33 (15.88) | 51.17 (16.53)
Statistical Analysis 1: Comparison: Cilostazol vs Placebo; Repeated ANOVA, tested for group*time interaction effect of ADCS-ADL scores on three data points (Baseline, 12-week, 24-week); Test type: Superiority or Other; p = 0.82, Repeated ANOVA

5. Secondary Outcome: Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB)
Description: Measured by professionally trained clinicians. Higher score indicates more severe AD symptoms.
  Score Scale: 0-18 (min-MAX)
Time Frame: Baseline, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 5.11 (2.30) | 4.72 (1.56)
  12-week | 5.42 (2.05) | 5.28 (2.18)
  24-week | 5.44 (2.49) | 5.33 (2.88)
Statistical Analysis 1: Comparison: Cilostazol vs Placebo; Repeated ANOVA, tested for group*time interaction effect of Summed CDR scores on three data points (Baseline, 12-week, 24-week); Test type: Superiority or Other; p = 0.79, Chi-squared

6. Secondary Outcome: Fazekas Scale
Description: Level of severity of white matter lesions in AD patients who can be legitimately administered with cilostazol. Measured by professionally trained clinicians.
  The higher score indicates more severe white matter lesion. Max-min: 0-3
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 18 | 18
participants
  Number of Patients Scored 1 | 13 | 11
  Number of Patients Scored 2 | 3 | 5
  Number of Patients Scored 3 | 2 | 2
Statistical Analysis 1: Comparison: Cilostazol vs Placebo; Distribution of Fazekas scale in two groups according to Chi-square test results; Test type: Superiority or Other; p = 0.87, Chi-squared

ADVERSE EVENTS:
Arm/Group | Cilostazol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/18 | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol (N=18) | Placebo (N=18)
Nausea, Dizziness (General disorders) | 1 (1) | 0 (0)
GI discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No